CLINICAL TRIAL: NCT00825006
Title: The Effects of Anodal Stimulation on Left Ventricular Desynchrony and Hemodynamics in Patients With a Biventricular Pacemaker
Brief Title: The Effects of Anodal Stimulation on Echocardiographic Outcome in Patients With Cardiac Resynchronization Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr Alon Barsheshet, Sheba Medical Center, Heart Institute
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-08-5076-MG-CTIL
Record Dates: First submitted 2008-03-09; First posted 2009-01-19 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronization therapy; Anodal stimulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Dual site pacing (LV tip electrode and RV tip electrode)
- Triple site pacing (Experimental): Triple site pacing(LV tip electrode,RV tip electrode and RV ring electrode)
  Interventions: Device: Triple site pacing mode

INTERVENTIONS:
Device: Triple site pacing mode — The experimental "Triple site pacing mode" includes pacing with Cardiac resynchronization therapy device using two leads; one in the right ventricle (RV) and one in the left ventricle (LV) but stimulates three sites: LV tip, RV tip and RV ring (instead of the usual two sites: LV tip and RV ring.
  Patients with evidence of improved LV dyssinchrony parameters during the triple pacing mode (anodal stimulation) will be programmed to anodal stimulation for 3 months.
  Other Names: anodal stimulation, triple site pacing
  Arms: Triple site pacing

SUMMARY:
To investigate the hemodynamic, inter and intraventricular desynchrony effects of anodal stimulation and triple site pacing compared with the usual dual site pacing by echocardiography and Tissue Doppler Imaging.

DETAILED DESCRIPTION:
Thirty patients who underwent CRT and had evidence of anodal stimulation will be included in the study. All patients undergo a conventional echocardiography after 10 minutes of continuous triple site pacing and after 10 minutes of continuous dual site pacing (Customary biventricular pacing).Echocardiography studies will be performed to measure dP/dT using continuous flow Doppler velocity profiles of mitral regurgitation, LV volumes and Left ventricular ejection fraction. Left intraventricular desynchrony is assessed by using TDI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biventricular pacemakers who met currently accepted indications for CRT, including dilated cardiomyopathy with LV ejection fraction < 35% (ischemic and nonischemic etiologies) with New York Heart Association class III to IV congestive heart failure and QRS duration > 120 ms.

Exclusion Criteria:

* Patients with first generation CRT device
* Integrated bipolar defibrillator device
* Atrial fibrillation during the screening phase
* Patients who cannot tolerate triple site pacing for several minutes (i.e diaphragmatic pacing)
* Patients with epicardial LV leads
* Patients with LV leads located out of the lateral or posterolateral areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial Performance Index, dP/dT | After 10 minutes of triple site pacing and 10 minutes of dual sute pacing

SECONDARY OUTCOMES:
Inter and intraventricular dyssynchrony parameters, LV volumes, LVEF | After 10 minutes of triple site pacing and 10 minutes of dual site pacing

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glikson, MD, Principal Investigator — Heart Institute, Sheba Medical Center
Locations (1):
- Heart Institute, Sheba Medical Center, Tel Litwinsky, Israel